CLINICAL TRIAL: NCT04993209
Title: Double-blind, Randomized, With an Active Control Vaccine, Phase I Clinical Trial for Evaluation of Safety and Immunogenicity of a Recombinant Inactivated COVID-19 Vaccine in Adults in Brazil - ADAPTCOV
Brief Title: Clinical Trial of the COVID-19 Vaccine (Recombinant, Inactivated) in Brazil
Acronym: ADAPTCOV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCV-01-IB
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Coronavirus Infections; Healthy
Keywords: Vaccine; SARS-CoV-2; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — NDV-HXP-S COVID-19 vaccine; sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Stage A (blinding form) will verify the product safety and support the decision on the dose selection among 1 μg, 3 μg and 10 μg, based on the immune response assessment. These results will also explore the response against 2 variants of concern in SARS-CoV-2: γ and β.
Who Masked: Participant, Care Provider, Investigator
Masking Description: An electronic central randomization system will be used to designate the investigational product (IP) that each participant must receive. A team study non-blind, qualified member (nurse/pharmacist) will obtain the corresponding randomization, will separate the respective IP, will blind the product and deliver it to blind staff. The product will be in a syringe that is in a blister labeled with the sponsor's name, IP code, administration route, IP dose and expiration date. The study non-blind staff will not have contact with the participants, will not have access to identification data or any other involvement with the study, besides randomizing the participant, separating the syringe containing placebo or vaccine, checking if the information on the blister label corresponds the information on the cartridge label and the syringe is labeled with the clinical trial code, ID, corresponding visit and investigator's name. Blinding is maintained with the opacity of the label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NDV-HXP-S 1μg (Experimental): NDV-HXP-S 1μg with an interval of 28 days apart. A dose escalation will be performed with an interval of two days between each dose in a blinded form. The aim is to verify the product safety and support the decision on the dose selection among three alternatives, 1 μg, 3 μg and 10 μg, based on the immune response evaluation. These results will also explore the response against two variants of concern in SARS-CoV-2: γ and β. The Phase I (former stage A) is designed as a non-inferiority test comparing the three different doses.
  Interventions: Biological: NDV-HXP-S 1μg
- NDV-HXP-S 3μg (Experimental): NDV-HXP-S 3μg with an interval of 28 days apart. A dose escalation will be performed with an interval of two days between each dose in a blinded form. The aim is to verify the product safety and support the decision on the dose selection among three alternatives, 1 μg, 3 μg and 10 μg, based on the immune response evaluation. These results will also explore the response against two variants of concern in SARS-CoV-2: γ and β. The Phase I (former stage A) is designed as a non-inferiority test comparing the three different doses.
  Interventions: Biological: NDV-HXP-S 3μg
- NDV-HXP-S 10μg (Experimental): NDV-HXP-S 10μg/0.5mL intramuscularly, with an interval of 28 days apart. A dose escalation will be performed with an interval of two days between each dose in a blinded form. The aim is to verify the product safety and support the decision on the dose selection among three alternatives, 1 μg, 3 μg and 10 μg, based on the immune response evaluation. These results will also explore the response against two variants of concern in SARS-CoV-2: γ and β. The Phase I (former stage A) is designed as a non-inferiority test comparing the three different doses.
  Interventions: Biological: NDV-HXP-S 10μg
- Adsorbed inactivated COVID-19 vaccine (CoronaVac) (Active Comparator): Adsorbed inactivated COVID-19 vaccine 600 SU dose (0.5 mL) with an interval of 28 days apart Intramuscular (deltoid). In the original version of protocol, the control arm consisted in placebo use. There was a changing post hoc to Adsorbed inactivated COVID-19 vaccine (CoronaVac) due to decision of Data and Safety Monitoring Board, when 219 (50% of original sample) subjects have already included in the study. Therefore, those who received a placebo at the first vaccine visit started to receive active control vaccine and those who were included from that moment forward received two doses of active control vaccine. The original study protocol provided for the inclusion of the placebo arm (10% of population of study), in order to serve as a control for safety evaluations and to assess the attack rate of natural infection to which participants will be exposed during the study.
  Interventions: Other: Adsorbed inactivated COVID-19 vaccine (CoronaVac)

INTERVENTIONS:
Biological: NDV-HXP-S 1μg — NDV-HXP-S 1μg 0.5mL 2 doses intramuscular (deltoid) 28 days apart
  Arms: NDV-HXP-S 1μg
Biological: NDV-HXP-S 3μg — NDV-HXP-S 3μg 0.5mL 2 doses intramuscular (deltoid) 28 days apart
  Arms: NDV-HXP-S 3μg
Biological: NDV-HXP-S 10μg — NDV-HXP-S 10μg 0.5mL 2 doses intramuscular (deltoid) 28 days apart
  Arms: NDV-HXP-S 10μg
Other: Adsorbed inactivated COVID-19 vaccine (CoronaVac) — Adsorbed inactivated COVID-19 vaccine 600 SU/0.5 mL 2 doses intramuscular (deltoid) 28 days apart
  Arms: Adsorbed inactivated COVID-19 vaccine (CoronaVac)

SUMMARY:
NDV-HXP-S is an inactivated COVID-19 vectored-vaccine virus using the Newcastle Disease Virus as basis and expressing S protein from SARS-CoV-2 stabilized in pre-fusion form with Hexapro technology.

This vaccine was successfully tested in non-clinical study with a good safety profile and eliciting neutralizing antibodies against SARS-CoV-2. Clinical testing is conducted by an international consortium including three different manufacturers. Butantan, in Brazil, is one of them.

DETAILED DESCRIPTION:
The present protocol aims, to respond to several regulatory requirements to advance the clinical development of the product through a dose-escalation, controlled, randomized, adult clinical trial. The results of the Phase I (former Stage A), allow us to base the decision to evaluate the safety and immunogenicity of three doses of HDV-HXP-S (1μg, 3μg or 10μg).

ELIGIBILITY:
Inclusion criteria

1. Adults aged between 18 and 59 years at the time of consent;
2. Agree to periodical contacts via phone, electronic means and home visits;
3. Good health conditions (absence of a clinically significant medical condition, acute or chronic, determined by medical history, physical examination, and clinical evaluation by the investigator);
4. Body Mass Index (BMI) of 17 to 40 kg/m² at the time of screening;
5. Intention of participating in the study by signing the Informed Consent Form;
6. A negative result for antibody testing against SARS-CoV-2 by CLIA performed within 7 days prior to study immunization;
7. No history of COVID-19 diagnosed by RT-PCR or antigen testing at screening visit and therefore within 72 hours prior to study enrollment;
8. No history of vaccination against COVID-19.

Exclusion criteria

1. Use any product under investigation within 90 days prior to randomization or plan to use a product during the period of participation in the study;
2. Have received vaccine in the last 28 days prior to inclusion in the study, or have immunization scheduled throughout the study period;
3. Evidences of uncontrolled active neurological, cardiac, pulmonary, hepatic or renal disease, according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
4. Have a history of severe allergic reaction or anaphylaxis to the vaccine or study vaccine components;
5. History of being allergic to chicken or eggs;
6. History of angioedema or anaphylactic reaction;
7. Have suspected or confirmed fever within 72 hours prior to vaccination or an axillary temperature above 37.8°C* on the day of vaccination (inclusion may be delayed until participant completes 72 hours without fever);
8. Altered vital signs, clinically relevant in the opinion of the principal investigator;
9. Neoplastic diseases (except basal cell carcinoma and cervical carcinoma in situ);
10. Suspected or confirmed diseases with compromised immune system including: congenital or acquired immunodeficiencies and uncontrolled autoimmune diseases according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
11. Make use of immunosuppressive therapies six months prior to inclusion in the study or schedule use of immunosuppressants within two years of inclusion in the study. The dose of corticosteroids considered immunosuppressive is the equivalent to prednisone at a dose of 2,0 mg/kg/day for adults, for more than a week. The continuous use of topical or nasal corticosteroids is not considered immunosuppressive. The following therapies are considered immunosuppressive: antineoplastic drugs, radiotherapy, immunosuppressants to induce tolerance to transplants, among others.
12. Have received blood products (transfusions or immunoglobulins) in the last three months prior to inclusion in the study, or schedule administration of blood products or immunoglobulins within two years of inclusion in the study.
13. Have a history of bleeding disorders (e.g., clotting factor deficiency, coagulopathy, platelet dysfunction), or prior history of significant bleeding or bruising after IM injection or venipuncture;
14. Have a history of any alcohol or drug abuse in the last 12 months prior to inclusion in the study that has caused medical, professional or family problems, as indicated by the clinical history;
15. Behavioral, cognitive, or psychiatric illness that, in the opinion of the principal investigator or medical representative, affects the participant's ability to understand and collaborate with the requirements of the study protocol;
16. The participant is a member of the team conducting the study or is in a dependent relationship with one of the members of the team conducting the study. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents), as well as employees or students who are directly dependent on the Researcher or local personnel conducting the study;
17. Any other condition that, in the opinion of the principal investigator or medical representative, may jeopardize the safety or rights of a potential participant or prevent them from complying with this protocol.
18. Abnormalities in screening laboratory tests considered to be exclusionary in the opinion of the principal investigator or medical representative. Grade 1 alterations are considered non-significant unless the principal investigator or medical representative indicates otherwise. If any alteration in the tests is considered temporary, the tests may be repeated in up to three opportunities during the screening period;
19. Positive serological tests for the human immunodeficiency virus (ELISA anti-HIV1/2); Hepatitis B (HbsAg or Anti-HBc) or Hepatitis C (total ELISA anti-HCV);

    For females:
20. Pregnancy (confirmed by a positive β-hCG test), breastfeeding and/or expressing intention to engage in sexual practices with reproductive potential without using a contraceptive method in the three months following vaccination

    * The temperature measured with a temporal thermometer is considered equivalent to the axillary temperature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse reactions. | 7 days after each vaccination.
  Number and intensity of solicited local and systemic adverse reactions.
Safety: Laboratory evaluations | 7 days after each vaccination.
  Number, severity and summary of clinically significant changes of hematological (hemoglobin [g/dL], white blood cells [cells/mm³] and platelets [count per mm³]) and biochemical evaluations (creatinine [mg/dL], AST [U/L], ALT [U/L], and total bilirubin [mg/dL]) since the baseline within 7 days after each vaccination.
Immunogenicity: Percentage of seroconversion. | 42(+7) days after the first dose.
  Percentage of positive SARS-CoV-2 pseudovirus neutralization assay in a participant with a baseline negative result (Wuhan strain).
Immunogenicity: Neutralization GMT SARS-CoV-2 pseudovirus. | 28 days after the first vaccination.
  Neutralization GMT against SARS-CoV-2 pseudovirus (Wuhan strain)
Immunogenicity: Neutralization GMT SARS-CoV-2 pseudovirus. | 14 days after the second vaccination.
  Neutralization GMT against SARS-CoV-2 pseudovirus (Wuhan strain)
Immunogenicity: Neutralization GMT SARS-CoV-2 pseudovirus. | 42(+7) days after the first dose.
  Neutralization GMT against SARS-CoV-2 pseudovirus (beta and gamma strains)

SECONDARY OUTCOMES:
Safety: all unsolicited adverse reactions. | 28 days after each vaccination.
  Number, intensity, and relatedness of all unsolicited adverse reactions.
Safety: serious and medically-attended adverse reactions. | Throughout the entire study period.
  Number, intensity, and relatedness of serious adverse reactions
Safety: events of special interest. | Throughout the entire study period.
  Number, intensity, and relatedness of events of special interest.
Immunogenicity: Levels of antibodies. | At baseline, 28 days after the first vaccination, and 14 days after the second vaccination, and 3, 6, 9, and 12 months after first vaccination.
  Levels of antibodies against SARS-CoV-2 Nucleocapsid protein and RBD
Immunogenicity: Neutralization GMT of SARS-CoV-2 pseudovirus. | 28 days after the first vaccination, and 14 days after the second vaccination.
  Neutralization GMT against SARS-CoV-2 pseudovirus per age group
Exploratory Endpoints: Levels of antibodies. | At baseline, 28 days after the first vaccination, and 14 days after the second vaccination, and 3 months, 6 months, 9 months, and 12 months after first vaccination.
  Levels of antibodies against SARS-CoV-2 Nucleocapsid protein and RBD.
Exploratory Endpoints: Neutralization GMT of SARS-CoV-2 pseudovirus. | at 3 months, 6 months, 9 months, and 12 months after first vaccination in subjects.
  Neutralization GMT against SARS-CoV-2 pseudovirus at 3 months, 6 months, 9 months, and 12 months after first vaccination in subjects.
Exploratory Endpoints - COVID-19 cases. | 14 days after first and second vaccination.
  Number and intensity of COVID-19 cases diagnosed.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Castro Boulos, MD,PhD, Study Director — Butantan Institute
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Peixoto de Miranda EJF, Calado RT, Boulos FC, de Sousa Moreira JA, Machado FF, Almeida MAALDS, Da Rocha MCO, Infante V, Mercer LD, Hjorth R, Scharf R, White J, Polyak C, Raghunandan R, Garcia-Sastre A, Sun W, Palese P, Krammer F, Innis B, Pereira CG, Kallas EG. Safety and immunogenicity of an inactivated recombinant Newcastle disease virus vaccine expressing SARS-CoV-2 spike: Results of a randomized vaccine-controlled phase I ADAPTCOV trial in Brazil. Vaccine. 2025 Apr 11;52:126680. doi: 10.1016/j.vaccine.2024.126680. Epub 2025 Mar 3. PMID 40037239